CLINICAL TRIAL: NCT05947487
Title: Phase I/II Study of CD70 Targeted CAR-T Cell Treatment in CD70 Positive Advanced/Metastatic Solid Tumors
Brief Title: CD70 Targeted CAR-T Cells in CD70 Positive Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-080
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumor, Adult
Keywords: CD70; advanced or metastatic
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD70-targeting CAR-T cells (Experimental): Enrolled participants will be given a preconditioning regimen consisted of albumin-bound paclitaxel, cyclophosphamide and fludarabine before the infusion of CD70-CAR-T cells.
  Enrolled patients in this arm will be administered CD70-CAR-T cells in 3+3 based escalation manner.
  Interventions: Biological: CD70-targeting CAR-T cells

INTERVENTIONS:
Biological: CD70-targeting CAR-T cells — Dose escalation:
  Dose1 (1×10^6 cells/kg) , Dose 2(3×10^6 cells/kg) ,Dose 3 (1×10^7cells/kg);
  Dose expansion: RP2D
  Drug: Albumin-bound paclitaxel
  Administered intravenously at dose of 100-200mg/m2 on day -5;
  Drug: Cyclophosphamide
  Administered intravenously at dose of 15-30mg/kg on day -3 and day -2;
  Drug: Fludarabine
  Administered intravenously at dose of 30mg/m2 on day -3 and day -2;

SUMMARY:
In this single-center, single-arm,prospective, open-label, phase 1/2 study, the safety and efficacy of autologous CD70 targeted chimeric antigen receptor modified T (CAR-T) cell therapy will be evaluated in patients with CD70 antigen positive advanced/metastatic solid tumors . In this clinical trial, at least 12 eligible patients in dose escalation period will be enrolled to receive 3 doses of CD70-CAR cell therapy according to the "3+3" principle. In dose expansion period, additional at most 21 eligible patients will be enrolled to receive CD70-CAR-T cell therapy at dose of recommended phase 2 dose(RP2D).

DETAILED DESCRIPTION:
Currently, CAR-T cell therapy has already achieved tremendous success in the treatment of hematological malignancies,however, it remains a severe challenge to treat solid tumors due to multiple obstacles,such as absence of tumor specific antigens, complex immunosuppressive tumor microenvironment, and tumor heterogeneity.

CD70 is a member of the tumor factor superfamily and has been found to be highly expressed on the surface of several solid and hematological tumors, correlating with inferior prognosis.Targeting CD70 has emerged as potential novel immunotherapeutic strategy. Investigators have developed CD70-CAR-T cells that could effectively expand and survive，producing strong anti-tumor effects in animal models. Based on the preclinical data, we conduct this clinical trial in order to test the the safety profiles and anti-tumor activities of CD70-CAR-T cells in vivo. In dose escalation period, at least 12 eligible patients will be enrolled and receive 3 doses of CD70-CAR-T cell therapy (1 × 10^6 cells/kg, 3 × 10^6 cells/kg, 1 × 10^7 cells/kg) according to the "3+3" principle. In dose expansion period, additional at most 21 eligible patients will be enrolled to receive CD70-CAR-T cell infusion at dose of RP2D, which is determined by data from dose escalation period, including occurrence of dose limiting toxicities (DLT), pharmacokinetics/pharmacodynamics, efficacy and other parameters, to furtherly evaluate the safety and efficacy profiles of CD70-CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. ECOG performance status ≤2 and Estimated life expectancy of more than 3 months.
3. Histopathological confirmed advanced or metastatic solid tumors failed to at least first-line treatment or initially diagnosed advanced/metastatic solid tumors that have no NCCN guideline recommended standard first-line therapy. CD70 antigen expression level ≥ 30%.
4. At least one measurable lesion at baseline per RECIST version 1.1.
5. Fresh solid tumor samples or formalin-fixed paraffin embedded tumor archival samples within 6 months are necessary; Fresh tumor samples are preferred. Subjects are willing to accept tumor rebiopsy in the process of this study.
6. Adequate organ function as defined by the following criteria: ANC≥1.5x10^9/L; Platelet count ≥75x10^9/L; Hemoglobin ≥90 g/L;Serum AST and serum ALT, ≤3.0 x ULN (≤5 x ULN for patients with liver cancer or metastases); Total serum bilirubin ≤1.5 x ULN(≤3 x ULN for patients with liver cancer or metastases); Serum creatinine ≤1.5 xULN or creatinine clearance of ≥60 mL/min.
7. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
8. Ability to understand and sign a written informed consent documen.

Exclusion Criteria:

1. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
2. Received cytotoxic chemicals, monoclonal antibodies, or immunotherapy within 4 weeks or 5 half-lives before enrollment;
3. Pregnant, lactating, or breastfeeding females;
4. Known positive test result for human immunodeficiency virus (HIV) oracquired immune deficiency syndrome (AIDS);Active infection of hepatitis B virus (HBV), or hepatitis C virus (HCV);
5. History of allergy or intolerance to study drug components;
6. Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation;
7. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
8. Known brain metastases or active central nervous system (CNS).Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
9. Previous or concurrent cancer within 5 years prior to treatment start except for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors;
10. Any serious underlying medical (eg, pulmonary, renal, hepatic,gastrointestinal, or neurological) or psychiatric condition or any issue that would limit compliance with study requirements;
11. Vaccination within 30 days of study enrollment;
12. Previously received CD70-CAR T cell therapy;
13. Being participating any other trials or withdraw within 4 weeks;
14. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | Up to 12 months since the initiation of CD70-CAR-T cell therapy.
  AE is defined as any adverse medical event from the date of randomization to 12 months after CD70-CAR-T cell infusion. Among them, CRS and ICANS were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Incidence of dose limiting toxicities (DLTs) | Up to 28 days since the initiation of CD70-CAR-T cell therapy
  DLT was defined as CD70-CAR-T cells-related events with onset within first 28 days following infusion: The development of Grade (G) 3 or higher grade CRS lasting > 2 weeks; All G4 non-hematologic toxicities.
Maximum tolerated dose (MTD) | Up to 28 days since the initiation of CD70-CAR-T cell therapy
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.

SECONDARY OUTCOMES:
Number and copy number of CD70-CAR-T cells | Up to 3 years
  Number and copy number of CD70-CAR-T cells are evaluated by number in peripheral blood and tumor tissue.
Objective response rate (ORR) | Up to 3 years
  Objective response rate includes complete response and partial response defined by investigators according to RECIST 1.1or iRECIST criteria.
Progression Free Survival (PFS) | Up to 3 years
  Progression Free Survival is defined as the time from the initiation of CD70-CAR-T cell therapy to documented disease progression or death.
Time to response (TTR) | Up to 3 years
  Time to response is defined as the time from the initiation of CD70-CAR-T cell therapy to first assessed CR or PR by investigators according to RECIST 1.1or iRECIST criteria.
Duration of response (DOR) | Up to 3 years
  Duration of response is defined as the time from objective response until documented tumor progression among responders.
Overall Survival (OS) | Up to 3 years
  Overall Survival is defined as the time from the initiation of CD70-CAR-T cell therapy to documented disease progression or death.
Pharmacodynamics: Peak level of cytokines in serum | Up to 28 days since the initiation of CD70-CAR-T cell therapy
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.

CONTACTS AND LOCATIONS:
Overall Officials: Yangbin Zhao, Ph.D, Study Director — UTC Therapeutics Inc.
Locations (1):
- China, Beijing, Iotherapeutic Department of Chinsese PLA Gereral Hospital, China